CLINICAL TRIAL: NCT05093881
Title: Long-term Follow-up of Patients With Alcoholic Liver Cirrhosis Who Had Administered Cellgram-LC in PMC-P-07 Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmicell Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PMC-P-07-01
Record Dates: First submitted 2021-10-13; First posted 2021-10-26 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Alcoholic Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Alcoholic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cellgram-LC (Experimental): Patients with Alcoholic Liver Cirrhosis who had administered Cellgram-LC in PMC-P-07 study.
  Interventions: Biological: Cellgram-LC

INTERVENTIONS:
Biological: Cellgram-LC — Patients who had administered Cellgram-LC in PMC-P-07 study

SUMMARY:
This Long-term follow-up is designed to evaluate the safety of patient with Alcoholic Liver Cirrhosis who had administered Cellgram-LC in PMC-P-07 study.

DETAILED DESCRIPTION:
To evaluate the safety for 60 months after a single dose of Cellgram-LC in patients with alcoholic liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. Those who participated in PMC-P-07 clinical trials and received Cellgram-LC
2. Those who voluntarily agreed in writing to participate in this investigation

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-24 (Actual); Primary Completion 2026-08-24 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of AESI | For 5 years
  death, neoplasms or malignancies in tissues or organs, Immune response including exacerbation or new outbreaks of previous autoimmune diseases, Other delayed AE related to Cellgram LC)
Rate of Liver transplant | For 5 years
  Liver transplant

CONTACTS AND LOCATIONS:
Overall Officials: Moonyoung Kim, Principal Investigator — Wonju Severance Christian Hospital
Locations (11):
- South Korea (11):
  - Soonchunhyang University Hospital, Bucheon-si
  - Soonchunhyang University Hospital, Cheonan
  - Gangwon National University Hospital, Chuncheon
  - Hallym Univ. Medical Center, Chuncheon
  - Gangneung Asan Hospital, Gangneung-si
  - Eunpyeong St. Mary's Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Soonchunhyang University Hospital, Seoul
  - Wonju Severance Christian Hospital, Wŏnju
  - Yongin Severance Hospital, Yŏngin